CLINICAL TRIAL: NCT06194383
Title: Optimization of the Treatment of Hyperpyrexia and Associated Symptoms in the Pediatric Emergency Department (FEVER_ED)
Brief Title: Treatment of Hyperpyrexia and in the Pediatric Emergency Department (FEVER_ED)
Acronym: FEVER_ED
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID6119; Fondazione Policlinico Univers (Other Grant/Funding Number: Fondazione Policlinico Universitario A. Gemelli IRCCS)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fever represents the main cause of admission to the emergency room in older people pediatric. It occurs in the presence of a wide range of pathologies, from infectious forms (the most common, viral or bacterial) up to more complex and/or systemic forms (such as inflammatory or neoplastic ones). The drugs currently indicated for the management of fever in children are: paracetamol and ibuprofen. There are no recent studies conducted in pediatric population, who have demonstrated the greater effectiveness of therapy with paracetamol or ibuprofen, The objective of our study is, therefore, to identify which therapy is most appropriate for controlling body temperature e of associated symptoms in pediatric patients arriving in the emergency room with fever.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (aged between 6 months 0 and 20 years)
* fever (T > 38°C) with/without associated symptoms, treated with standard antipyretic drugs orally (paracetamol, ibuprofen or paracetamol/ibuprofen combination)
* who have expressed their consent to participate in the study.

Exclusion Criteria:

* age <6 months or >20 years;
* patients who did not express consent to participate in the study

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (aged between 6 months 0 and 20 years), with fever (T > 38°C) with/without associated symptoms, treated with standard antipyretic drugs orally (paracetamol, ibuprofen or paracetamol/ibuprofen combination)
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Response to the treatment as evaluation of associated symptoms | 1 hour
  Evaluation of associated symptoms by pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy